CLINICAL TRIAL: NCT00559468
Title: A Multi -Center, Randomized, Parallel Group, Safety Assessor Blinded Trial Comparing Efficacy and Safety of 4.0 mg.Kg-1 Sugammadex , Administered at T1 3-10% After Continuous Infusion of Rocuronium, and Pharmacokinetics of Rocuronium, Between Subjects Receiving Maintenance Anesthesia Using Propofol and Subjects Receiving Maintenance Anesthesia Using Sevoflurane
Brief Title: Sugammadex After Continuous Infusion of Rocuronium During Sevoflurane and Propofol Anesthesia (P05949; MK-8616-028)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05949; 19.4.312 (Other: Organon Protocol Number); MK-8616-028 (Other: Merck Protocol Number); 2006-004072-12 (Other: EudraCT Number)
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Rocuronium; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex + Sevoflurane (Experimental): After receiving sevoflurane and the last dose of rocuronium, at the reappearance of first twitch (T1; 3-10% starting amplitude), a dose of 4.0 mg/kg sugammadex was administered.
  Interventions: Drug: Sugammadex; Drug: Rocuronium; Drug: Sevoflurane
- Sugammadex + Propofol (Experimental): After receiving propofol and the last dose of rocuronium, at the reappearance of first twitch (T1; 3-10% starting amplitude), a dose of 4.0 mg/kg sugammadex was administered.
  Interventions: Drug: Sugammadex; Drug: Rocuronium; Drug: Propofol

INTERVENTIONS:
Drug: Sugammadex — Single dose 4.0 mg/kg sugammadex, administered at T1 3-10% after continuous infusion of rocuronium
  Other Names: Org 25969; MK-8616
Drug: Rocuronium — Single bolus dose 0.6 mg/kg rocuronium and continuous infusion rocuronium
  Other Names: Esmeron®; Rocuronium Bromide
Drug: Sevoflurane — Sevoflurane IV administered for induction and maintenance of anesthesia, based on randomization.
  Other Names: Ultane®
  Arms: Sugammadex + Sevoflurane
Drug: Propofol — Propofol IV administered for induction and maintenance of anesthesia, based on randomization.
  Other Names: Diprivan®
  Arms: Sugammadex + Propofol

SUMMARY:
The objective of the trial was to show equivalence in recovery from neuromuscular block after a single dose of 4.0 mg/kg sugammadex, administered at first twitch (T1) 3-10% after continuous infusion of rocuronium, between participants receiving maintenance anesthesia using propofol and participants receiving sevoflurane, to investigate the safety and to compare the plasma levels of rocuronium in participants after continuous infusion of rocuronium and before the administration of sugammadex, under either propofol or sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 20 years but under 65 years of age;
* Participants of American Society of Anesthesiologists (ASA) class 1-3;
* Participants scheduled for a surgical procedure under general anesthesia requiring neuromuscular relaxation with the use of a neuromuscular blocking agent (NMBA) with an anticipated duration of surgery between 2 and 5 hours;
* Participants scheduled for a surgical procedure in supine position;
* Participants who had given written informed consent.

Exclusion Criteria:

* Participants in whom difficult intubation was expected because of anatomical malformations;
* Participants known or suspected to have neuromuscular disorders affecting NMB and/or significant renal dysfunction. In Germany, this also included serum creatinine and blood urea nitrogen outside local reference ranges;
* Participants known or suspected to have a (family) history of malignant hyperthermia;
* Participants known or suspected to have an allergy to medications used during general anesthesia;
* Participants receiving medication interfering with NMBAs, such as antibiotics, anticonvulsants and Mg^2+; based on the dose and time of administration;
* Pregnant or lactating females;
* Female participants of childbearing potential not using any birth control or using only hormonal contraception as birth control;
* Participants who had already participated in trial CT 19.4.312, or in another trial with sugammadex;
* Participants who had participated in another clinical trial, not pre-approved by Organon, within 30 days of entering into CT 19.4.312.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-12-07 (Actual); Primary Completion 2007-03-02 (Actual); Study Completion 2007-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Rex C, Wagner S, Spies C, Scholz J, Rietbergen H, Heeringa M, Wulf H. Reversal of neuromuscular blockade by sugammadex after continuous infusion of rocuronium in patients randomized to sevoflurane or propofol maintenance anesthesia. Anesthesiology. 2009 Jul;111(1):30-5. doi: 10.1097/ALN.0b013e3181a51cb0. PMID 19512873
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had a surgical procedure using a general anesthesia (with sevoflurane or propofol) and rocuronium for endotracheal intubation and maintenance of neuromuscular block (NMB) were enrolled in this study.
Pre-assignment Details: Out of 52 randomized participants, 51 received treatment.
Period: Overall Study
Arm/Group | Sugammadex + Sevoflurane | Sugammadex + Propofol
Started | 26 | 26
Treated | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all randomized participants receiving study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex + Sevoflurane | Sugammadex + Propofol | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (12.4) | 50.4 (8.3) | 50.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Time From Start Administration of Sugammadex to Recovery of Fourth Twitch/First Twitch (T4/T1) Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive Train of Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 ratio (expressed as a decimal from 0 [loss of T4] up to 1.0 [no NMB]) indicates the extent of recovery from NMB. In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: Up to 3 minutes after sugammadex administration
Population: All randomized participants who received sugammadex and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex + Sevoflurane | Sugammadex + Propofol
Number analyzed (Participants) | 26 | 25
minutes | 1.45 (0.45) | 1.32 (0.40)

2. Secondary Outcome: Mean Time From Start of Administration of Sugammadex to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 ratio (expressed as a decimal from 0 [loss of T4] up to 1.0 [no NMB]) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: Up to 3 minutes after sugammadex administration
Population: All randomized participants who received sugammadex and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex + Sevoflurane | Sugammadex + Propofol
Number analyzed (Participants) | 26 | 25
minutes | 1.07 (0.25) | 1.02 (0.28)

3. Secondary Outcome: Mean Time From Start of Administration of Sugammadex to Recovery of the T4/T1 Ratio to 0.8
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 ratio (expressed as a decimal from 0 [loss of T4] up to 1.0 [no NMB]) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: Up to 3 minutes after sugammadex administration
Population: All randomized participants who received sugammadex and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex + Sevoflurane | Sugammadex + Propofol
Number analyzed (Participants) | 26 | 25
minutes | 1.20 (0.35) | 1.12 (0.30)

ADVERSE EVENTS:
Time Frame: Up to 7 days after sugammadex treatment
Description: All randomized participants receiving study treatment are included.
Arm/Group | Sugammadex + Sevoflurane | Sugammadex + Propofol
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 21/26 | 21/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex + Sevoflurane (N=26) | Sugammadex + Propofol (N=25)
Constipation (Gastrointestinal disorders) | 12 (12) | 5 (5)
Flatulence (Gastrointestinal disorders) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 9 (11) | 5 (6)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Impaired healing (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 14 (14) | 19 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (9) | 2 (2)
Sleep disorder (Psychiatric disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognizes the right of the investigators to publish, but all publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.